CLINICAL TRIAL: NCT05675553
Title: A Randomized Controlled Trial Protocol Testing the Efficacy of Robot-Assisted Intelligent Rehabilitation Treatment in Patients With Alcohol Use Disorders
Brief Title: The Efficacy of Robot-Assisted Intelligent Rehabilitation Treatment in Patients With AUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MZhao-011
Record Dates: First submitted 2022-12-28; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot-assisted rehabilitation intelligent treatment (Experimental): Both groups will receive treatment as usual(TAU) provided by the clinical team, including medication, exercise, and psychotherapy. Robot-assisted intelligent rehabilitation treatment will be delivered to participants in the testing group through an addiction prevention and relapse intervention intelligent system.
  Interventions: Device: robot-assisted rehabilitation intelligent treatment; Other: treatment as usual
- treatment as usual (Other): Participants in the treatment-as-usual group were offered standard treatment at the mental health hospitals, which consisted of group and/or individual therapy, as determined by the clinical team.
  Interventions: Other: treatment as usual

INTERVENTIONS:
Device: robot-assisted rehabilitation intelligent treatment — Participants assigned to this condition were offered 10 individual sessions of robot-assisted rehabilitation treatment, delivered by the Robot-assisted rehabilitation intelligent system. The system contains 10 core cognitive-behavioral therapy (CBT) skill topics (such as functional analysis, coping skills training, reviewing practice exercises, and explaining CBT concepts). A robot therapist demonstrates the target CBT skills and assigns homework to participants. The treatment framework is semi-structured through human-computer interaction. The forms of interaction include inquiries, statements, recommendations summaries, and knowledge assessments.
  Arms: robot-assisted rehabilitation intelligent treatment
Other: treatment as usual — Both groups will receive treatment as usual, including medication, exercise, and psychological education.

SUMMARY:
We aimed to test the efficacy of robot-assisted intelligent rehabilitation treatment in patients with alcohol use disorders with a randomized controlled trial. Specifically, the objective of this trial is to determine whether the robot-assisted intelligent rehabilitation treatment plus treatment as usual has greater efficacy than traditional therapy in the treatment of alcohol use disorders.

DETAILED DESCRIPTION:
Based on artificial intelligence technology, face recognition technology, and virtual reality technology to develop an available Robot-assisted rehabilitation intelligent system. Then, using this intelligent system as a new way of Psychotherapy to provide treatment for patients with alcohol use disorders, and compare with traditional treatment to verify the efficacy and safety of the Robot-assisted rehabilitation intelligent system in Chinese patients with alcohol use disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-55;
2. Meeting DSM-5 criteria for alcohol use disorders;
3. Withdrawing alcohol for less than 12 months;
4. Ability to use computers;
5. Signing informed consent;

Exclusion Criteria:

1. Having comorbidities of other neuropsychiatric diseases;
2. Diseases that affect cognitive function, such as a history of head trauma, cerebrovascular disease, epilepsy, etc.
3. With a family history of mental illness
4. Not familiar with computer operation, unable to complete assessment and treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Desire for alcohol | 3 months
  The primary outcome is patients' desire for alcohol,measured by Visual Analogue Scale(VAS).

SECONDARY OUTCOMES:
Change Readiness and Treatment Eagerness | 3 months
  The secondary outcome includes participants' Change Readiness and Treatment Eagerness, measured by the Stages of Change Readiness and Treatment Eagerness Scale(SOCRATES).
Impulsiveness | 3 months
  The secondary outcome includes participants' level of impulsiveness, measured by the Barratt Impulsiveness Scale(Barratt).
Anxiety | 3 months
  The secondary outcome includes the participants' level of anxiety, measured by generalized Anxiety Disorder-7(GAD-7).
Depression | 3 months
  The secondary outcome includes the participants' level of depression, measured by Patient Health Questionnaire-9(PHQ-9).
Perception of stress | 3 months
  The secondary outcome includes participants' perception of stress, measured by the Perceived Stress Scale(PSS).
Sleep Quality | 3 months
  The secondary outcome includes participants' sleep quality, measured by Pittsburgh Sleep Quality Index(PSQI).
coping style | 3 months
  The secondary outcome includes participants' coping style, measured by Simplified Coping Style Questionnaire(SCSQ).
use of alcohol | 3 months
  The secondary outcome includes participants' use of alcohol.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No